CLINICAL TRIAL: NCT05878132
Title: 'Smart Reminder': a Feasibility Pilot Study on the Effects of a Wearable Device Treatment on the Hemiplegic Upper Limb in Persons With Stroke
Brief Title: 'Smart Reminder': a Feasibility Pilot Study on the Effects of a Wearable Device Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Kenneth N. K. Fong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20220704001
Record Dates: First submitted 2023-04-03; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: Stroke; telerehabilitation; Wearable device; Upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single-blinded randomized crossover trial
Who Masked: Outcomes Assessor
Masking Description: Randomization was stratified based on the participant's baseline upper limb severity according to the FTHUE-HK. Masking to treatment allocation for therapist and participants was not feasible.
  Only the outcome assessor was blinded to the treatment allocation and participants were instructed not to tell the assessor their group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wearable device group (Experimental): Participants in the experimental group will be instructed to wear the wristwatch device five days per week for a minimum of 3 hours per day and engage in telerehabilitation, 1hour per day for 5 times per week over 4 weeks. Weekly, there will be a 30-minute therapy consultation.
  Interventions: Device: Wearable device -'Smart Reminder'
- Conventional therapy group (Active Comparator): The participants in the conventional group will receive similar in-home upper limb exercises as the wearable device group, with the prescribed exercises presented in the form of a pictorial handout rather than an in-app video. They are instructed to perform the exercises 1hour per day, 5times per week over 4 weeks. Weekly, there will be a 30-minute therapy consultation.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Device: Wearable device -'Smart Reminder' — The wearable device, a wristwatch, has a Bluetooth function to link to mobile devices for the participants to view the prescribed videos and engage in telerehabilitation. It has sensors to monitor arm movements and provides multiple feedbacks (auditory, visual and tactile). Participants were instructed to practice the prescribed exercises -tailored according to the severity of UL paresis for the recommended therapy dose. The device recorded the angles of arm movement and the number of repetitions completed and data collected is uploaded to an encrypted cloud server for remote monitoring. Weekly, the participants will receive a 30-minute consultation session to review their progress and modify prescribed exercises based on the wearable device data.
  Arms: Wearable device group
Other: Conventional therapy — The participants in the control group received similar in-home upper limb exercises as the wearable device group, with the prescribed exercises presented in the form of a pictorial handout rather than an in-app video. They were instructed to perform the exercises for the recommended therapy dose and received a weekly therapy consultation as well. To monitor the participant's exercise compliance, they were instructed to record their daily exercise progress in the exercise log.
  Arms: Conventional therapy group

SUMMARY:
This pilot study examines the feasibility and potential effects on upper limb (UL) motor function using a wearable device integrated with a telerehabilitation function in the home setting with chronic stroke survivors.

The study seeks to address the question:

- Is wearable device intervention more effective in promoting arm recovery in stroke survivors than conventional therapy for home-based training? We hypothesize that using a multimodal feedback system in the wearable device can provide more effective training to improve the hemiplegic UL function of chronic stroke survivors than conventional therapy.

This is a single-blinded randomized crossover pilot trial. Twelve participants will be randomly assigned into two groups: the experimental (wristwatch) and the control (conventional therapy) groups. Participants in the experimental group will undergo a 4-week wearable device treatment followed by a 4-week conventional training.

Participants in the control group will complete conventional therapy and then wearable device treatment. There will be a 3-week washout period between treatments. Upper limb motor outcome measures will be evaluated at the following intervals: baseline, post-treatment at 4-week, after a 3-week washout period for pre-intervention, and post-intervention after crossover by research assistants blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* unilateral hemispherical involvement
* diagnosis of stroke with onset ≥ three months
* hemiplegic upper limb with Functional test for hemiplegic upper extremity-Hong Kong version (FTHUE-HK) ≥ score of 3 (maximum of 7) (Fong et al., 2004).
* no complaint of excessive pain and swelling over the hemiplegic arm
* able to provide informed consent to participate.

Exclusion Criteria:

* participating in another similar form of experimental study during the same period
* having a history of botulinum toxin injection in the past three months
* having other significant upper limb impairment, i.e. fixed contractures, frozen shoulder, and severe arthritis
* having a diagnosis which would interfere in the use of the device, i.e. visual impairment, active cardiac issues and palliative treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Fugl Meyer Upper Extremity assessment | Change from baseline at 4 weeks
  The FMA-UE is a 3-point scale with a maximum score of 66 that measures the synergistic pattern and ability to make arm movements.The total score is further subdivided into upper-extremity and hand subscores with a total score of 66 (Fugl Meyer et al., 1975)
Change from preintervention at 7-week (after crossover) Fugl Meyer Upper Extremity assessment | Change from 7-week at 11 weeks
  The FMA-UE is a 3-point scale with a maximum score of 66 that measures the synergistic pattern and ability to make arm movements.The total score is further subdivided into upper-extremity and hand subscores with a total score of 66 (Fugl Meyer et al., 1975)
Change from baseline Motor Activity Log (MAL) | Change from baseline at 4 weeks
  The MAL is a self-reported questionnaire designed to assess how frequently and effectively patients utilize their affected arm daily. It consists of 2 subscales to measure patients' perceived amount of arm use (MAL-AOU) and quality of arm use (MAL-QOM) (Uswatte, Taub, Morris, Light & Thompson, 2006)
Change from preintervention at 7-week (after crossover) Motor Activity Log (MAL) | Change from 7-week at 11 weeks
  The MAL is a self-reported questionnaire designed to assess how frequently and effectively patients utilize their affected arm daily. It consists of 2 subscales to measure patients' perceived amount of arm use (MAL-AOU) and quality of arm use (MAL-QOM) (Uswatte, Taub, Morris, Light & Thompson, 2006)
Change from baseline Action Research Arm Test | Change from baseline at 4 weeks
  The ARAT is a frequently used assessment tool to assess hemiplegic upper limb function. It consists of 19 items comprising four domains: grasp, grip, pinch, and gross motor, and has a total score of 57 (Lyle, 1981).
Change from preintervention at 7-week (after crossover) Action Research Arm Test | Change from 7-week at 11 weeks
  The ARAT is a frequently used assessment tool to assess hemiplegic upper limb function. It consists of 19 items comprising four domains: grasp, grip, pinch, and gross motor, and has a total score of 57 (Lyle, 1981).
Change from baseline Active range of motion (AROM) of shoulder and elbow | Change from baseline at 4 weeks
  The active ROM of the shoulder (flexion) and elbow (flexion/ extension) will be evaluated using a manual goniometer.
Change from preintervention at 7-week (after crossover) Active range of motion (AROM) of shoulder and elbow | Change from 7-week at 11 weeks
  The active ROM of the shoulder (flexion) and elbow (flexion/ extension) will be evaluated using a manual goniometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Kenneth FONG, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fong, K., Ng, B., Chan, D., Chan, E., Ma, D., Au, B., ... & Occupational Therapy Central Coordinating Committee. (2004). Development of the Hong Kong version of the functional test for the hemiplegic upper extremity (FTHUE-HK). Hong Kong Journal of Occupational Therapy, 14(1), 21-29.
- [Background] Lyle RC. A performance test for assessment of upper limb function in physical rehabilitation treatment and research. Int J Rehabil Res. 1981;4(4):483-92. doi: 10.1097/00004356-198112000-00001. No abstract available. PMID 7333761
- [Background] Uswatte G, Taub E, Morris D, Light K, Thompson PA. The Motor Activity Log-28: assessing daily use of the hemiparetic arm after stroke. Neurology. 2006 Oct 10;67(7):1189-94. doi: 10.1212/01.wnl.0000238164.90657.c2. PMID 17030751
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616